CLINICAL TRIAL: NCT03527849
Title: The Effect of Mindfulness-Based Stress Reduction on Pain and Function in Persons With Knee Osteoarthritis
Brief Title: Effects of Mindfulness-Based Stress Reduction on Knee Osteoarthritis
Acronym: MBSR on KOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1180036
Record Dates: First submitted 2018-04-20; First posted 2018-05-17 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Knee Osteoarthritis; Knee Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Mindfulness-Based Stress Reduction; Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study will be structured as a parallel-group controlled trial. The Principal Investigator will assign participants into the three groups. This will allow for equalization of distribution of participants across the three groups. It will not be possible to blind the participants to which arm of the trial they are participating in, as the content or lack thereof of their activities will be obvious to them. For results analysis, collaborators at the UCD West Coast Metabolomics Center will be blinded to the treatment of the respective samples, thus eliminating potential bias during analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-Person MBSR Course (Experimental)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Online MBSR Course (Experimental)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- In-Person HEP (Active Comparator)
  Interventions: Behavioral: Health Enhancement Program

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — The intervention will be an MBSR course.
  Other Names: Mindfulness
  Arms: In-Person MBSR Course; Online MBSR Course
Behavioral: Health Enhancement Program — Propose to use an active control training, the Health Enhancement Program (HEP), an intervention designed to isolate mindfulness as a testable active ingredient. HEP and MBSR are structurally equivalent in that they share the same amount of in- and out-of class work time. The content of the HEP intervention meet the following criteria: (1) class activities match MBSR activities as closely as possible, (2) activities represent valid, active, therapeutic ingredients in their own right, and (3) these ingredients do not include mindfulness.
  Other Names: HEP
  Arms: In-Person HEP

SUMMARY:
The purpose of this study is to see if stress reduction can lead to less pain due to knee osteoarthritis. To do this the investigators will compare two types of stress reduction modalities, Mindfulness-Based Stressed Reduction (MBSR) and a Health Enhancement Program (HEP). Both include stress reduction techniques, but MBSR has a mindfulness component that includes meditation. MBSR will be provided either in-person or online and HEP will be in-person. The assignment to the stress reduction program will be determined by the Principal Investigator. In order to assess for stress reduction and pain reduction the investigators will use validated measuring tools before, during, and after the course instructions.

DETAILED DESCRIPTION:
The current study is aiming to compare two stress reduction programs in order to see if stress reduction may lead to less pain due to knee osteoarthritis (OA). There are two stress reduction programs being compared, Mindfulness-Based Stress Reduction (MBSR) and a Health Enhancement Program (HEP). MBSR is a secular program that trains mindfulness meditation for stress reduction and to increase emotional regulation skills. It is defined as "paying attention in a particular way, on purpose, in the present moment, and non-judgmentally." Mindfulness refers to a set of meditation practices that develop a wide array of cognitive skills which include: attention regulation, response inhibition, and emotion regulation. HEP is an educational course intended to teach participants about their disease, factors influencing disease progression, nutrition, physical activity including walking and stretching, and functional movement. Key difference between these two is MBSR includes the mindfulness component, and MBSR will be taught either in-person or online. HEP will only consist of an in-person course.

The online MBSR course will be offered through: http://www.breathworks-mindfulness.org.uk/mindfulness-for-health. The investigators propose to use an active control training, the Health Enhancement Program (HEP), an intervention designed to isolate mindfulness as a testable active ingredient.

The duration of an individual subject's participation in the study will be at least 10 weeks starting from the screening visit all the way to the follow-up visit.

The in-person MBSR course consists of 8 weekly classes plus one all-day class between Weeks 6 and 7, and is sequential. Depending on when a participant is consented, they may have to wait until a new 8-week course is available in order to begin. The HEP course also consists of 8 weekly classes and will start when a group of 7-10 participants have been assigned to the HEP intervention. The online MBSR course is designed to last 8 weeks and can be started at any time.

Since initiation of the in-person MBSR or HEP courses will depend upon when subjects are enrolled, it is not possible to provide the maximum length of time for a subject's participation. However long the subject's participation, they are only expected to complete 2 in-clinic visits and 8 weeks of class (plus 1 all-day class for MBSR).

Weekly classes are 2.5 hours with the one-day retreat lasting from 10am to 5pm on a weekend day. The online MBSR course is roughly 20 minutes per day for 6-7 days of the week for 8 weeks.

HEP and MBSR are structurally equivalent, both using a group format that meets once a week for 2.5 hours for 8 weeks, plus home participation, but the in-person MBSR includes an "all day" component after week 6. The content of the HEP intervention meets the following criteria: (1) class activities match MBSR activities as closely as possible, (2) activities represent valid, active, therapeutic ingredients in their own right, and (3) these ingredients do not include mindfulness.

All participants will be assigned into one of the three courses by the Principal Investigator. Prior to the initial class of the participants' respective course, blood will be collected, and within two weeks after the final class, participants will return to collect the second set of blood samples. These collections prior and after treatment will be at the clinic, visits to the clinic may last from 1 to 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Positive "Frequent Knee Pain" question
* Radiographically confirmed knee OA (Kellgren/Lawrence ≥ 2)

Exclusion Criteria:

* Scheduled to have knee replacement surgery within 6 months from enrollment
* Rheumatoid arthritis or another inflammatory arthritis
* Known avascular necrosis (death of bone due to lack of blood supply)
* Failure to comply with run-in procedures: poor attendance or non-compliant with completing the activity
* Major psychiatric illness, cognitive impairment or alcohol/substance abuse
* Non-English speaking

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | At First Clinical Visit (Baseline Week 1), During Treatment (Once per week for 8 Weeks), at Second Clinical Visit (Post-Treatment Week 10), this will be done through the participant's duration in the study on average lasting 10 weeks.
  A joint specific questionnaire used to measure the condition of patients with knee osteoarthritis, pain, stiffness, and physical functioning of the inflicted joints. Each question is answered by selecting a box from a scale of 0-10 (0=No Pain, 10=Extreme Pain). The investigators plan on collecting a baseline measurement prior to the treatment, weekly measurements through the treatment (1 per week for 8 weeks), and another after the treatment is completed to track changes.

SECONDARY OUTCOMES:
Change in Emotion Regulation Questionnaire (ERQ) | At First Clinical Visit (Baseline Week 1), Mid-Treatment (Week 5), at Second Clinical Visit (Post-TreatmentWeek 10), this will be done through the participant's duration in the study on average lasting 10 weeks.
  A self-reported questionnaire that identifies the habitual use of two emotional regulation strategies, between cognitive reappraisal and expressive suppression.
  Answered in a scale ranging from 1-7 (1=strongly disagree, 4=neutral, 7=strongly agree). Answered prior to receiving treatment, half-way through treatment completion, and post-treatment.
Change in 5 Facet Mindfulness Questionnaire (FFMQ) | At First Clinical Visit (Baseline Week 1), Mid-Treatment (Week 5), at Second Clinical Visit (Post-Treatment Week 10), this will be done through the participant's duration in the study on average lasting 10 weeks.
  A self-reported questionnaire intended to measure the five factors to conceptually be involved with mindfulness. It is answered using a 1-5 scale (1=never or very rarely true, 2=rarely true, 3=sometimes true, 4=often true, 5=very often or always true). Answered prior to receiving treatment, half-way through treatment completion, and post-treatment.
Change in Pain Catastrophizing Scale (PCS) | At First Clinical Visit (Baseline Week 1), Mid-Treatment (Week 5), at Second Clinical Visit (Post-Treatment Week 10), this will be done through the participant's duration in the study on average lasting 10 weeks.
  A self-reported questionnaire used to quantify an individual's pain experience through a series of questions asking about the individual's feelings and thoughts about when they are in pain.
  Answered in a scale of 0-4 (0=not at all, 1=to a slight degree, 2=to a moderate degree, 3=to a great degree, 4=all the time). Answered prior to receiving treatment, half-way through treatment completion, and post-treatment.
Change in Plasma Cortisol Levels | At First Clinical Visit (Baseline Week 1) and at Second Clinical Visit (Post-Treatment Week 10)
  Cortisol is a hormone the human body releases in times of stress. Because the investigators are aiming to reduce stress the investigative team will be collecting blood (4mL RED-top Vacutainer tube) prior to beginning treatment (respective stress reduction course) and after the course is completed to assess if there were changes in cortisol levels. Cortisol levels will be obtained in micrograms per deciliter (ug/dL).
Change in Cytokine Plasma Levels | At First Clinical Visit (Baseline Week 1) and at Second Clinical Visit (Post-Treatment Week 10)
  Cytokines are markers secreted by cells that help direct cell function during an immune response. The investigators will collect blood and process serum for analysis to measure and track changes in cytokine levels responsible for inflammation. The blood will be collected at the first clinical visit and the second clinical visit. The measurements will be interpreted in picograms per milliliter (pg/mL).
Change in Oxylipin Plasma Levels | At First Clinical Visit (Baseline Week 1) and at Second Clinical Visit (Post-Treatment Week 10)
  Oxylipin inflammation markers will be measured from plasma processed from collected blood at the first and second clinical visits. There are usually 84 markers and are positively detected and quantified even in healthy individuals using 150uL of plasma. The investigative team expects there to be higher concentrations of these markers in elderly subjects with OA pain, furthermore, the investigators expect differences in concentrations of these markers for the different treatments. These values will be addressed in nanomolar (nM).

CONTACTS AND LOCATIONS:
Overall Officials: Barton L. Wise, Principal Investigator — UC Davis School of Medicine; Philippe Goldin, Principal Investigator — UC Davis Betty Irene School of Nursing
Locations (1):
- University of California, Davis Medical Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan on making unidentifiable participant data for all primary and secondary outcome measures available. No information linking the data to the individual participant will be released, but measurements, averages, and statistical analysis will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available 6 months after study completion.
Access Criteria: Data access requests will be reviewed by Principle Investigators.

REFERENCES:
- [Background] Kabat-Zinn J, University of Massachusetts Medical Center/Worcester. Stress Reduction Clinic. Full catastrophe living: using the wisdom of your body and mind to face stress, pain, and illness. New York, N.Y.:Delacorte Press; 1990.
- [Result] Trelle S, Reichenbach S, Wandel S, Hildebrand P, Tschannen B, Villiger PM, Egger M, Juni P. Cardiovascular safety of non-steroidal anti-inflammatory drugs: network meta-analysis. BMJ. 2011 Jan 11;342:c7086. doi: 10.1136/bmj.c7086. PMID 21224324
- [Result] Wolfe MM, Lichtenstein DR, Singh G. Gastrointestinal toxicity of nonsteroidal antiinflammatory drugs. N Engl J Med. 1999 Jun 17;340(24):1888-99. doi: 10.1056/NEJM199906173402407. No abstract available. PMID 10369853
- [Result] Abou-Raya S, Abou-Raya A, Helmii M. Duloxetine for the management of pain in older adults with knee osteoarthritis: randomised placebo-controlled trial. Age Ageing. 2012 Sep;41(5):646-52. doi: 10.1093/ageing/afs072. Epub 2012 Jun 27. PMID 22743149
- [Result] Chappell AS, Desaiah D, Liu-Seifert H, Zhang S, Skljarevski V, Belenkov Y, Brown JP. A double-blind, randomized, placebo-controlled study of the efficacy and safety of duloxetine for the treatment of chronic pain due to osteoarthritis of the knee. Pain Pract. 2011 Jan-Feb;11(1):33-41. doi: 10.1111/j.1533-2500.2010.00401.x. PMID 20602715
- [Result] Wise BL, Niu J, Zhang Y, Wang N, Jordan JM, Choy E, Hunter DJ. Psychological factors and their relation to osteoarthritis pain. Osteoarthritis Cartilage. 2010 Jul;18(7):883-7. doi: 10.1016/j.joca.2009.11.016. Epub 2010 Mar 24. PMID 20346403
- [Result] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Result] Hilton L, Hempel S, Ewing BA, Apaydin E, Xenakis L, Newberry S, Colaiaco B, Maher AR, Shanman RM, Sorbero ME, Maglione MA. Mindfulness Meditation for Chronic Pain: Systematic Review and Meta-analysis. Ann Behav Med. 2017 Apr;51(2):199-213. doi: 10.1007/s12160-016-9844-2. PMID 27658913
- [Result] O'Leary K, O'Neill S, Dockray S. A systematic review of the effects of mindfulness interventions on cortisol. J Health Psychol. 2016 Sep;21(9):2108-21. doi: 10.1177/1359105315569095. Epub 2015 Feb 10. PMID 25673371
- [Result] Rosenkranz MA, Lutz A, Perlman DM, Bachhuber DR, Schuyler BS, MacCoon DG, Davidson RJ. Reduced stress and inflammatory responsiveness in experienced meditators compared to a matched healthy control group. Psychoneuroendocrinology. 2016 Jun;68:117-25. doi: 10.1016/j.psyneuen.2016.02.013. Epub 2016 Feb 20. PMID 26970711
- [Result] Yadav RK, Magan D, Mehta N, Sharma R, Mahapatra SC. Efficacy of a short-term yoga-based lifestyle intervention in reducing stress and inflammation: preliminary results. J Altern Complement Med. 2012 Jul;18(7):662-7. doi: 10.1089/acm.2011.0265. PMID 22830969
- [Result] MacCoon DG, Imel ZE, Rosenkranz MA, Sheftel JG, Weng HY, Sullivan JC, Bonus KA, Stoney CM, Salomons TV, Davidson RJ, Lutz A. The validation of an active control intervention for Mindfulness Based Stress Reduction (MBSR). Behav Res Ther. 2012 Jan;50(1):3-12. doi: 10.1016/j.brat.2011.10.011. Epub 2011 Nov 11. PMID 22137364
- [Result] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Result] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Result] Lange T, Vansteelandt S, Bekaert M. A simple unified approach for estimating natural direct and indirect effects. Am J Epidemiol. 2012 Aug 1;176(3):190-5. doi: 10.1093/aje/kwr525. Epub 2012 Jul 10. PMID 22781427

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/49/NCT03527849/Prot_SAP_000.pdf